CLINICAL TRIAL: NCT03112200
Title: A Randomized Controlled Trial of the Subchondroplasty® Procedure With Arthroscopy Versus Arthroscopy Alone for Treatment of Bone Marrow Lesions in the Knee
Brief Title: Subchondroplasty® Knee RCT
Acronym: PRESERVE Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: MedNet Solutions (Unknown); Medical Metrics Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KC.CR.I.AM.16.1
Record Dates: First submitted 2017-03-27; First posted 2017-04-13 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Bone Marrow Edema; Knee Pain Chronic; Knee Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis
Keywords: Subchondroplasty; Arthroscopy; Bone Substitute Material; Subchondral Bone Defect; AccuFill; Bone Marrow Lesion; Knee Replacement; Knee Replacement Alternative
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Arthroscopy

STUDY DESIGN:
Intervention Model Description: A stratified blocked randomization will be used to assign subjects to either Subchondroplasty with arthroscopy or to arthroscopy alone in a 2:1 ratio. Individual sets of blocks will be determined within study site and lesion polarity status (unipolar vs. bipolar).
Who Masked: Participant
Masking Description: The surgeon will be blinded to the treatment group until the time of surgery to avoid potential selection bias during the screening process. The subject will be blinded to the treatment group. The research coordinator will consult the central randomization list to determine which group the subject is in. Subjects may be randomized prior to surgery to allow for OR set-up. However, randomization should be performed as close to the time of surgery as possible to reduce the risk of randomization failures due to cancelled procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Subchondroplasty with Arthroscopy (Active Comparator): After randomization to the study group, subjects assigned to the Subchondroplasty + Arthroscopy group will undergo the Subchondroplasty portion of the procedure before or after the Arthroscopy portion per the surgeon's discretion. All operative procedures are to be performed under aseptic conditions according to the institution's standards.
  Interventions: Procedure: Subchondroplasty with Arthroscopy
- Arthroscopy Alone (Sham Comparator): After randomization, subjects assigned to the Arthroscopy control group will undergo arthroscopy of the study knee with one or more of the following procedures:
  * Partial meniscectomy
  * Lavage
  * Debridement
  * Loose body removal
  * Synovectomy
  * Removal of osteophytes in the notch or locations other than those adjacent to BML(s)
  Superficial skin incision(s) should be created at the typical AccuPort® access point(s) as if the subject had undergone Subchondroplasty. The incisions should be closed in the typical fashion.
  Interventions: Procedure: Arthroscopy Alone

INTERVENTIONS:
Procedure: Subchondroplasty with Arthroscopy — The Subchondroplasty® (SCP®) Procedure targets and fills bone defects with AccuFill® Bone Substitute Material utilizing an arthroscopic / percutaneous approach. Using intraoperative fluoroscopy, the bone defect is localized relative to MRI findings The appropriate AccuPort® Delivery Cannula is drilled to the bone defect. AccuFill® Bone Substitute Material is then injected into the subchondral bone defect. The calcium phosphate (CaP) fills the edematous void and hardens within the Bone Marrow Lesion. The CaP is resorbed over time and replaced with new bone during the healing process.
  Arms: Subchondroplasty with Arthroscopy
Procedure: Arthroscopy Alone — An endoscopic examination, therapy and surgery of the knee joint.
  Arms: Arthroscopy Alone

SUMMARY:
This is a multi-center, prospective, single-blinded, two-arm study, randomized to include approximately 134 subjects treated with Subchondroplasty (SCP) + Arthroscopy and 67 subjects with arthroscopy alone.

The primary objective of this study is to demonstrate superiority of Subchondroplasty with arthroscopy compared to arthroscopy alone for treatment of Bone Marrow Lesions (BMLs) in the knee.

DETAILED DESCRIPTION:
This is a multicenter, prospective, single-blinded, two-arm, randomized study. Enrolled subjects will have a single Bone Marrow Lesion of the tibia, single BML of the femur, or adjoining Bone Marrow Lesions of tibia and femur. Subjects will also be surgical candidates for knee arthroscopy due to mechanical symptoms, meniscus tear, loose body and/or synovitis.

A stratified blocked randomization will be used to assign subjects to either Subchondroplasty with arthroscopy or to arthroscopy alone in a 2:1 ratio. Individual sets of blocks will be determined within study site and lesion polarity status (unipolar vs. bipolar).

Subjects will be enrolled within 60 days prior to surgery and take part in follow-up visits for two years following surgery. A preoperative visit will occur at the time of enrollment. Follow-up visits were to initially occur at the study site at 6 weeks, 3 months, 6 months, 12 months, and 24 months post-surgery. Telephone follow-up interviews to be be performed at 9 and 18 months post-surgery. Target enrollment was 201 subjects, to include 134 subjects in the treatment group (Subchondroplasty + Arthroscopy) and 67 subjects in the control group (Arthroscopy alone).

As of October 2020, follow-up has been amended to be completed remotely, where all visits can be performed electronically and/or via telephone.

Subjects will complete the study at the 24 month follow-up visit. For the purposes of this protocol, a revision will be defined as any partial or total joint arthroplasty or any bone fixation, bone grafting or bone substitute procedure in the same compartment in the study knee.

ELIGIBILITY:
Inclusion Criteria:

* Candidates must meet ALL of the following:

  1. Voluntary signature of the Institutional Review Board/Research Ethics Board approved Informed Consent,
  2. Male or female subjects between the ages of 30 to 75 years,
  3. Body Mass Index ≤ 40 (BMI=kg/m2),
  4. Has experienced pain in study knee for at least 3 months,
  5. Kellgren-Lawrence grade 1-3 Osteoarthritis, as reviewed on preoperative XR imaging, in the study knee,
  6. BML is confirmed on T2 weighted or Proton Density MR Imaging by presence of white signal,
  7. Single BML of tibia, single BML of femur, or adjoining BML's of tibia & femur, in the same compartment, extending to the articular surface of the joint,
  8. Surgical candidate for knee arthroscopy due to mechanical symptoms, meniscus tear, loose body and/or synovitis,
  9. Must record a response, at the preoperative study visit, of moderate to extreme pain for any one of the KOOS Pain Scale questions, P2 through P9,
  10. Index knee alignment is defined radiographically as one of the following: Neutral, ≤ 6° mechanical varus, or ≤ 6° mechanical valgus,
  11. Ligaments in the study knee are stable,
  12. The contralateral (non-study) knee is stable and functional,
  13. Is refractory to conservative non-surgical management

      1. having failed 2 or more of the following: hyaluronic acid injection, corticosteroid injection, NSAIDs, physical therapy, bracing, activity modification, or minimal surgical intervention (e.g., arthroscopy, debridement/chondroplasty, and/or loose body removal)
      2. and is ≥ 3 months from the start of treatment,
  14. Must be physically and mentally willing and able, in the Investigator's opinion at the time of enrollment, to be compliant with the protocol - including all follow-up visits, survey completion, weight-bearing restrictions, and post-operative rehabilitation.

Exclusion Criteria:

* Candidates will be excluded if they meet ANY of the following:

  1. BML caused by acute trauma less than 3 months prior to enrollment,
  2. Clinical and/or radiographic disease diagnosis of the index knee that includes any of the following:

     1. Kellgren-Lawrence Grade 4 Osteoarthritis with complete loss of joint space (bone-on-bone) or subchondral bone collapse,
     2. Rheumatoid arthritis, or history of septic or reactive arthritis,
     3. Gout or a history of gout or pseudogout in the affected knee,
     4. Has more than two clinically relevant BMLs in the index knee,
     5. Osteochondritis dissecans of the knee with significant bone loss,
     6. Collapse of subchondral bone,
     7. Clinically relevant BML located at ACL/PCL insertion,
     8. MRI evidence of frank ligament instability,
  3. Passive knee flexion < 110° or flexion contracture >30°,
  4. History of systemic diseases which could contribute to secondary arthropathies (e.g., sickle cell disease, hemochromatosis, or autoimmune disease),
  5. Has a neuromuscular, neurosensory, or musculoskeletal deficiency that limits the ability to perform objective functional assessment of either knee,
  6. If diabetic, blood glucose over 200 mg/dL at time of enrollment,
  7. Current daily tobacco or high nicotine product user or < 3 months from nicotine cessation,
  8. Presents a high surgical risk due to unstable cardiac and/or pulmonary disease,
  9. Has HIV or other immunodeficient state including subjects on immunosuppressant therapies, or has significant illness (metastasis of any type) that decreases the probability of survival to the 2 year endpoint,
  10. Is at substantial risk for the need of organ transplantation, such as renal insufficiency,
  11. Is pregnant or breast-feeding at the time of surgery,
  12. Has a history of any invasive malignancy (except non-melanoma skin cancer), unless treated with curative intent and with no clinical signs or symptoms of the malignancy for 5 years,
  13. Has primary bone tumor in the knee area,
  14. Anticipates having a lower extremity surgery other than the investigational surgery during the course of the study,
  15. Is participating concurrently in another clinical trial, or has participated in a clinical trial within 30 days of surgery,
  16. Is receiving prescription pain medication other than NSAIDs or acetaminophen for conditions unrelated to the index knee condition, chronic use of anticoagulants, or taking corticosteroids,
  17. Active joint infection or history of chronic joint infection at the surgical site,
  18. Prior total meniscectomy of index knee,
  19. Has primarily patellofemoral symptoms,
  20. Is indicated for concomitant procedures (i.e., microfracture, subchondral drilling, cartilage allograft, ligament or tendon repair, distal realignment/osteotomy, root repair) in the index knee, with the exception of incidental loose body removal, debridement, synovectomy, osteophyte removal in locations other than adjacent to BMLs, and/or partial meniscectomy,
  21. Has contraindications for Magnetic Resonance Imaging (MRI),
  22. Is receiving worker's compensation or is currently involved in litigation relating to the index knee,
  23. Has a history of substance abuse.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Composite Clinical Success | Superiority will be statistically tested at month 12 at p<0.01
  The primary objective of this study is to determine whether Subchondroplasty with arthroscopy is superior to arthroscopy alone for treatment of bone marrow lesions in the knee.
  Superiority will be evaluated in terms of Composite Clinical Success (CCS) requiring freedom from subsequent secondary surgical intervention (SSSI) and among those free from SSSI, a clinically meaningful reduction in self-reported pain based on a validated measure of subject-reported pain (improvement in KOOS (Knee Injury and Osteoarthritis Outcome Score) pain of at least 10 points at 12 months) .
  For the purpose of this study, SSSI will include any partial or total joint arthroplasty or any bone grafting or bone substitute procedure in the study knee.

SECONDARY OUTCOMES:
Change from baseline KOOS subscale scores at 12 Months | 12 months post-surgery
  Comparison of mean change in KOOS subscale scores (Pain, Activities of Daily Living), Symptoms, Sports and Recreation, Quality of Life)
Change from baseline Numeric Pain Score at 12 Months | 12 months post-surgery
  Comparison of mean Numeric Pain Score
Change from baseline EQ-5D score at 12 Months | 12 months post-surgery
  Comparison of mean EQ-5D score
Change from baseline Global Satisfaction score at 12 Months | 12 months post-surgery
  Comparison of mean Global Satisfaction score
Change from baseline x-rays to 12 Months | 12 months post-surgery
  X-ray evaluation of joint space narrowing, osteophyte and cyst formation and subchondral sclerosis
MRI analysis | 12 months post-surgery
  MRI analysis of bone marrow lesion variables
Incidence of post-operative complications and adverse events | 12 months post-surgery
  Incidence of post-operative complications and adverse events
Time to resolution of post-operative complications and adverse events | 12 months post-surgery
  Time to resolution of post-operative complications and adverse events
Incidence of joint injections | 12 months post-surgery
  Incidence of joint injections
Time to joint injections | 12 months post-surgery
  Time to joint injections
Incidence of re-operations and revisions | 12 months post-surgery
  Incidence of re-operations and revisions
Time to re-operations and revisions | 12 months post-surgery
  Time to re-operations and revisions
Healthcare utilization | 12 months post-surgery
  Estimated total healthcare expenditure through 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jason Dragoo, MD, Principal Investigator — University of Colorado, Denver
Locations (13):
- United States (12):
  - CORE Orthopaedic Medical Center, Encinitas, California
  - Loma Linda University Health System, Loma Linda, California
  - Stanford University, Stanford, California
  - Foundation for Orthopaedic Research and Education, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - MedStar Health Research Institute, Timonium, Maryland
  - New Mexico Orthopaedic Fellowship Foundation, Albuquerque, New Mexico
  - The Ohio State University, Columbus, Ohio
  - Hawkins Foundation, Greenville, South Carolina
  - Orthopedic Associates of Central Texas, Austin, Texas
  - University of Virginia, Charlottesville, Virginia
- Research St. Joseph's - Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No